CLINICAL TRIAL: NCT07355400
Title: Clinical Evaluation of the NeoPill Device for Reduction of Oral Bacterial Load in Patients With Fixed Orthodontic Appliances
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neofunction d.o.o. (Industry)
Collaborators: German Oncology Center, Cyprus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ЕЕВК/ЕП/2025/72
Record Dates: First submitted 2025-12-16; First posted 2026-01-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Dental Plaque
Keywords: Dental plaque; Oral bacterial load; Orthodontic appliances; Oral hygiene device; Mechanical oral cleaning
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Intervention Model Description: This is a single-arm, pre-post interventional study in which all participants receive a single standardized 30-second application of the NeoPill device. Oral bacterial load is assessed before and immediately after the intervention using paired oral swab samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NeoPill Device Intervention (Experimental): Participants in this single-arm study receive a single standardized 30-second application of the NeoPill oral hygiene device. Oral swab samples are collected immediately before and after device use to assess changes in aerobic bacterial load.
  Interventions: Device: NeoPill Oral Hygiene Device

INTERVENTIONS:
Device: NeoPill Oral Hygiene Device — The NeoPill is a reusable, battery-operated oral hygiene device applied intraorally for a standardized duration of 30 seconds. In this study, the device is applied once by trained study personnel. The intervention involves no chemical agents and no systemic exposure. The device is used to mechanically clean the oral cavity prior to post-intervention oral swab collection.

SUMMARY:
This study evaluates the effectiveness of the NeoPill oral hygiene device in reducing oral bacterial load in adults wearing fixed orthodontic appliances. Maintaining oral hygiene is challenging for orthodontic patients due to limited access around brackets and wires, and current solutions often rely on chemical-based products and disposable tools.

NeoPill is a reusable, battery-operated oral device designed to provide mechanical cleansing of the oral cavity. In this single-arm clinical evaluation, participants will undergo oral swab sampling before and immediately after a single 30-second application of the NeoPill device. The primary outcome is the change in aerobic bacterial load, measured as colony-forming units (CFUs), between pre- and post-treatment samples.

Participants will also complete a short questionnaire to assess usability, comfort, and overall experience with the device. The study aims to generate preliminary clinical and user-experience data to support further development of the NeoPill device.

DETAILED DESCRIPTION:
This is a single-arm, pre-post interventional clinical evaluation designed to assess the effectiveness of the NeoPill device in reducing aerobic bacterial load in the oral cavity of adults with fixed orthodontic appliances. The study will be conducted at the German Medical Institute in Limassol, Cyprus, and will enroll approximately 15 to 20 participants aged 18 years or older.

Eligible participants must be currently wearing fixed orthodontic appliances and able to provide informed consent. Exclusion criteria include recent antibiotic use, active oral infections, immunocompromised status, or systemic conditions that may affect oral flora.

After providing written informed consent, participants will undergo baseline oral swab collection from gingival areas and around orthodontic brackets on the upper second premolars. A trained research technician or nurse will then apply the NeoPill device for a standardized duration of 30 seconds, ensuring consistent positioning and technique across participants. Immediately following device application, a second oral swab will be collected from the same anatomical sites.

Both swab samples will be transported under controlled conditions to an accredited microbiology laboratory at the German Medical Institute, where aerobic culturing will be performed to quantify colony-forming units (CFUs). The primary outcome measure is the difference in CFU counts between pre- and post-intervention samples. Statistical analysis will be conducted using a Wilcoxon Signed Rank Test with a significance threshold of p < 0.05.

Following sample collection, participants will complete a structured questionnaire assessing comfort, usability, perceived experience, and willingness to use the NeoPill device regularly. Questionnaire data and laboratory results will be linked using study-specific identifiers and stored securely within a GDPR-compliant digital platform.

The study involves minimal risk to participants, limited primarily to temporary discomfort during swab collection or device use. No chemical agents or systemic interventions are involved. All data will be pseudonymised prior to analysis, and only anonymised results will be shared with the device manufacturer.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Currently wearing fixed orthodontic appliances
* Able and willing to provide written informed consent
* Able to comply with study procedures during a single study visit

Exclusion Criteria:

* Use of systemic antibiotics within the past 2 weeks
* Presence of active oral infections
* Known immunocompromised status
* Presence of systemic medical conditions that may affect oral bacterial flora

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2026-02-13 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Change in aerobic oral bacterial load | Immediately before and immediately after the intervention (same study visit)
  Difference in aerobic bacterial colony-forming unit (CFU) counts measured from oral swab samples collected immediately before and immediately after a single 30-second application of the NeoPill device.

SECONDARY OUTCOMES:
Participant-reported usability and comfort of the NeoPill device | Immediately after device use (same study visit)
  Participant-reported usability and comfort are assessed using a NeoPill Participant Usability and Comfort Questionnaire, a structured, study-specific survey administered immediately after device use.
  The composite usability score is derived from Likert-scale items assessing overall experience, discomfort/pain, and likelihood of future use.
  - Overall experience is rated on a 5-point Likert scale ranging from 1 (Very Unpleasant) to 5 (Very Pleasant).
  Higher scores indicate a more positive user experience.
  - Discomfort or pain during device use is rated on a 5-point Likert scale ranging from 1 (No Pain) to 5 (Severe Pain).
  Higher scores indicate greater discomfort.
  - Likelihood of regular future use is rated on a 5-point Likert scale ranging from 1 (Very Unlikely) to 5 (Very Likely).
  Higher scores indicate greater acceptability and usability.
  Responses are combined descriptively to evaluate overall usability and comfort of the NeoPill device.

CONTACTS AND LOCATIONS:
Overall Officials: Constantinos Zamboglou, Study Director — GMIC
Locations (1):
- German Medical Institute, Limassol, Cyprus

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because all study data are pseudonymised and analysed for the specific purposes defined in the study protocol and ethics approval, with no provision for secondary data sharing.